CLINICAL TRIAL: NCT03863366
Title: The Effect of a Single Dose of Prucalopride on Emotional Processing in Healthy Volunteers
Brief Title: Effects of Acute Prucalopride Administration in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Principal Investigator, drsusannahmurphy, Senior Research Fellow, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Acute_pruc
Record Dates: First submitted 2019-02-26; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Molecular Mechanisms of Pharmacological Action; Depression; Depressive Disorder; Mood Disorders; Mental Disorder; Antidepressive Agents; Cognition
Keywords: 5-HT4; Prucalopride; Resolor; Emotional Processing; Healthy Volunteers
MeSH Terms: conditions — Depression; Depressive Disorder; Mood Disorders; Mental Disorders | interventions — prucalopride

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to one of two groups (prucalopride or placebo). Participants in the prucalopride group will receive 1mg of the drug. Participants in the placebo group will receive a lactose placebo. Note that the study is not assessing the safety or efficacy of prucalopride, rather it is using prucalopride to assess the behavioural and neural effects of 5-HT4 partial agonists.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prucalopride (Experimental): 1mg prucalopride capsule
  Interventions: Drug: Prucalopride
- Placebo (Placebo Comparator): Lactose placebo capsule
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Prucalopride — 1mg prucalopride tablet, encapsulated in white capsule
  Other Names: Resolor
  Arms: Prucalopride
Other: Placebo — Lactose placebo tablet, encapsulated in white capsule
  Arms: Placebo

SUMMARY:
This study will investigate whether administration of a single dose of the serotonin receptor subtype 4 (5-HT4) partial agonist prucalopride has effects on emotional processing and non-emotional cognition in healthy volunteers, compared to placebo administration. Using an experimental medicine approach, the effects of prucalopride on cognitive biomarkers of antidepressant action will be characterised. In a double-blind design, participants will be randomised to receive a single dose of either prucalopride (1mg) or placebo. All participants will come for a Screening Visit to ensure their suitability for the study. If they meet study criteria, they will be invited to a Research Visit, where they will receive the study medication and wait for two hours while the drug reaches peak levels. After two hours they will be asked to complete a series of computer-based tasks measuring emotional, non-emotional cognitive processing, and reward processing. The primary study hypothesis is that acute prucalopride administration will have positive effects on processing facial expressions of emotion. Secondary hypotheses are that acute prucalopride administration will affect other measures of emotional processing, and non-emotional cognition.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 18-40 years
* Willing and able to give informed consent for participation in the study
* Sufficiently fluent English to understand and complete the task

Exclusion Criteria:

* Current usage of psychoactive medication (except the contraceptive pill, the Depo-Provera injection or the progesterone implant)
* Any past or current Axis 1 DSM-IV psychiatric disorder
* Significant medical condition
* Current or past gastro-intestinal disorder or irritable bowel syndrome
* Current pregnancy or breastfeeding
* Known lactate deficiency or any other problem absorbing lactose, galactose or glucose
* Current or past history of drug or alcohol dependency
* Participation in a psychological or medical study involving the use of medication within the last 3 months
* Previous participation in a study using the same, or similar, emotional processing tasks
* Smoker > 5 cigarettes per day
* Typically drinks > 6 caffeinated drinks per day

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2017-08-08 (Actual); Study Completion 2017-08-08 (Actual)

PRIMARY OUTCOMES:
Recognition of positive and negative facial expressions | Day 1: 2-5 hours post drug administration
  Accuracy to identify positive vs. negative facial expressions of emotion on the FERT

SECONDARY OUTCOMES:
Recall of emotional words | Day 1: 2-5 hours post drug administration
  Number of positive and negative words correctly (and incorrectly) recalled in the EREC task
Recognition of emotional words | Day 1: 2-5 hours post drug administration
  Number of positive and negative words correctly (and incorrectly) recognised in the EMEM task
Attentional vigilance to emotional faces | Day 1: 2-5 hours post drug administration
  Attentional vigilance to fearful and happy faces in the FDOT task
Recall of words Auditory Verbal Learning Task (AVLT) | Day 1: 2-5 hours post drug administration
  Number of items correctly and incorrectly recalled across blocks
Reward and loss sensitivity | Day 1: 2-5 hours post drug administration
  Proportion of participants on each trial that chose the correct (high probability) symbol in the win condition, and the incorrect (high probability) symbol in the loss condition of the PILT task
Working memory performance | Day 1: 2-5 hours post drug administration
  Mean accuracy and reaction time on 1-back, 2-back and 3-back conditions compared with 0-back condition on the N-back task
Contextual learning | Day 1: 2-5 hours post drug administration
  Difference between reaction time and accuracy on novel and repeated arrays in the contextual cueing task

CONTACTS AND LOCATIONS:
Overall Officials: Susannah E Murphy, DPhil, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Psychopharmacology and Emotion Research Laboratory — http://www.perloxford.org